CLINICAL TRIAL: NCT03213574
Title: Impact of Goal Directed Fluid Therapy in Robot-assisted Laparoscopic Urological Surgery for Low to Moderate Risk Patients
Brief Title: Impact of GDT in Robot-assisted Laparoscopic Urological Surgery for Low to Moderate Risk Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator is making changes to the protocol.
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Ronak Raval, MD, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5170073
Record Dates: First submitted 2017-02-06; First posted 2017-07-11 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Vascular Hypotension; Hypovolemia; Hypervolemia
Keywords: Goal directed fluid therapy
MeSH Terms: conditions — Hypotension; Hypovolemia; Edema | interventions — Control Groups

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): The control group will be administered intraoperative fluids throughout his or her surgery per the discretion of the anesthesiologist as is typical for this type of case. They will use an arterial line but without a FloTrac and therefore will have no data regarding the SVV.
  Interventions: Other: Control Group
- Treatment Group (Experimental): The treatment group will receive a FloTrac arterial line that will allow the anesthesiologist to administer intraoperative fluids based on the study algorithm.
  Interventions: Other: Treatment Group

INTERVENTIONS:
Other: Control Group — Intraoperative fluids will be administer per the discretion of anesthesia provider and not per SVV data or study protocol.
  Arms: Control Group
Other: Treatment Group — FloTrac arterial line data will be used to administer fluid bolus, based on study algorithm.
  Arms: Treatment Group

SUMMARY:
Robot assisted urological procedures are often long surgical cases that can potentially result in complicated postoperative hospital course. The amount of intravenous (IV) fluids administered to patients during these operations fluctuates based on the length of the case, surgical blood loss, hemodynamic monitors, and the discretion of the anesthesiologist. The goal of intraoperative fluid therapy is to maintain optimal tissue perfusion without causing fluid overload. We plan to use a goal directed fluid therapy protocol to optimize fluid status and analyze post-operative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing robot-assisted laparoscopic urological procedures in which the patient would have an arterial catheter placed as part of their routine inoperative anesthetic management

Exclusion Criteria:

* Age less than 18;
* current pregnancy;
* history of congestive heart failure, arrhythmias, coagulopathy, cerebral vascular disease , COPD, significant liver or renal impairment, required FloTrac per treating anesthesiologist;
* patient refusal to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Postoperative ileus | Up to 3 weeks postoperatively
  Time postoperatively to first bowel movement

SECONDARY OUTCOMES:
Acute kidney injury | Up to 3 weeks postoperatively
  Will be measured using the KDIGO criteria (UOP and Cr)
Respiratory compromise | Up to 3 weeks postoperatively
  Patients that require oxygen or invasive/non-invasive mechanical ventilation postoperatively
Need for diuresis | Up to 3 weeks postoperatively
  Use of a diuretic medication (ex. lasix, metolazone)
Hospital length of stay | Up to 4 weeks postoperatively
  Duration of stay in the hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No